CLINICAL TRIAL: NCT03844464
Title: Special Investigation for LORBRENA Tablets
Brief Title: Safety and Efficacy of Lorbrena
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7461018; NCT03844464 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2019-02-15; First posted 2019-02-18 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the following matters under post-marketing use of Lorbrena in patients who received this drug

1. Factors affecting the onset of central nervous system disorder
2. Effect of Lorbrena in combination with CYP3A inducers on the onset of hepatic dysfunction

ELIGIBILITY:
Inclusion Criteria:

* All administered patients

Exclusion Criteria:

* Nothing

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 683 patients
Sampling Method: Probability Sample
Enrollment: 1290 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions of central nervous system disorder and hepatic dysfunction | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- 3-22-7, Yoyogi, Shibuya-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461018